CLINICAL TRIAL: NCT02914795
Title: Platelet Function in Resuscitated Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 27-290ex14/15
Record Dates: First submitted 2016-05-12; First posted 2016-09-26 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non-resuscitated myocardial infarction: diagnostic analysis of platelet function of a matched historical cohort of the ATLANTIS-ACS trial
  Interventions: Other: diagnostic analysis of platelet function
- resuscitated myocardial infarction: diagnostic analysis of platelet function of the patient cohort included according to the inclusion criteria
  Interventions: Other: diagnostic analysis of platelet function

INTERVENTIONS:
Other: diagnostic analysis of platelet function — analysis of platelet aggregation using optical measurements as well as the commercial VerifyNow technique

SUMMARY:
Approx. 65% of resuscitated patients at the intensive care unit for internal medicine are due to myocardial infarction. Almost all patients are initially diagnosed and treated in the cath lab. Therapy usually consists of one or more stent implantations. After implantation of a coronary stent, dual platelet inhibition is necessary for 12 months. Insufficient platelet inhibition causes an pronounced increase in risk of stent thrombosis. Therefore, knowledge of the individual platelet function is valuable.

Several factors potentially promote a delayed or reduced mode of action of platelet function inhibitors in resuscitated patients:

1. oral administration is impossible and medication needs to be administered via a gastric line.
2. gastric absorption is delayed after resuscitation
3. according to current guidelines patients are treated with therapeutic hypothermia. Including the time of rewarming cooling period is ~48h

DETAILED DESCRIPTION:
Patients after successful resuscitation associated to a myocardial infarction will be included into the study the morning after the index event. Patients get dual platelet inhibition at the discretion of the interventionist. Patients are treated with therapeutic hypothermia according to the local Standard operating procedure for 24h and rewarming is performed within an additional 20h. Platelet function is measured every morning and Aspirin mediated as well as P2Y12 (purinergic G protein-coupled receptors-12)-inhibition mediated platelet function inhibition is recorded. All relevant clinical data including APACHE (Acute Physiology and Chronic Health Evaluation) and SOFA ( Sequential Organ Failure Assessment score) scores are collected.

The degree of platelet inhibition over time (7 days) and differences between the three drugs tested will be evaluated by optical aggregometry and by using the commercial VerifyNow test system.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction
* dual platelet inhibition
* resuscitation
* therapeutic hypothermia

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients surviving the first night after resuscitation due to myocardial infarction
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk von Lewinski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNicol A, Israels SJ. Platelets and anti-platelet therapy. J Pharmacol Sci. 2003 Dec;93(4):381-96. doi: 10.1254/jphs.93.381. PMID 14737006
- [Background] Tendera M, Wojakowski W. Role of antiplatelet drugs in the prevention of cardiovascular events. Thromb Res. 2003 Jun 15;110(5-6):355-9. doi: 10.1016/j.thromres.2003.08.003. PMID 14592562
- [Background] Gurbel PA, Bliden KP, Hiatt BL, O'Connor CM. Clopidogrel for coronary stenting: response variability, drug resistance, and the effect of pretreatment platelet reactivity. Circulation. 2003 Jun 17;107(23):2908-13. doi: 10.1161/01.CIR.0000072771.11429.83. Epub 2003 Jun 9. PMID 12796140
- [Background] Puri KS, Suresh KR, Gogtay NJ, Thatte UM. Declaration of Helsinki, 2008: implications for stakeholders in research. J Postgrad Med. 2009 Apr-Jun;55(2):131-4. doi: 10.4103/0022-3859.52846. PMID 19550060
- [Background] Siller-Matula JM, Lang I, Christ G, Jilma B. Calcium-channel blockers reduce the antiplatelet effect of clopidogrel. J Am Coll Cardiol. 2008 Nov 4;52(19):1557-63. doi: 10.1016/j.jacc.2008.07.055. PMID 19007592
- [Derived] Pruller F, Bis L, Milke OL, Fruhwald F, Patzold S, Altmanninger-Sock S, Siller-Matula J, von Lewinski F, Ablasser K, Sacherer M, von Lewinski D. Cangrelor Induces More Potent Platelet Inhibition without Increasing Bleeding in Resuscitated Patients. J Clin Med. 2018 Nov 15;7(11):442. doi: 10.3390/jcm7110442. PMID 30445678

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-resuscitated Myocardial Infarction | Resuscitated Myocardial Infarction
Started | 77 | 22
Completed | 77 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-resuscitated Myocardial Infarction | Resuscitated Myocardial Infarction | Total
Number analyzed (Participants) | 77 | 22 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 13 | 52
  >=65 years | 38 | 9 | 47
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.3 [59.3 to 72.7] | 65 [50 to 75.8] | 64.5 [60.5 to 72.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 3 | 21
  Male | 59 | 19 | 78
Region of Enrollment [Number; unit: participants]
  Austria | 77 | 22 | 99
Collagen AUC day 1 [Median (Inter-Quartile Range); unit: AU*min] — Aspirin reactivity was monitored by inducing platelet aggregation with 2 µg/mL collagen and 0.5 mmol L-1 arachidonic acid (AA, Chronolog Corp., Havertown, PA, USA), respectively.
  First measurement was on day one and thus represents baseline.
  AU*min | 219 [80.5 to 334.5] | 69.5 [46.7 to 195.6] | 185.8 [77 to 244]

OUTCOME MEASURES:

1. Primary Outcome: Platelet Inhibition Measured With Optical Aggregometry
Description: Median (Inter-Quartile Range) Collagen AUC values on Day 3 measured with optical aggregometry The more light signal is detected, the better thrombocyte function is.
Time Frame: day 3
Measure: Median (Inter-Quartile Range); unit: AU*min
Groups:
- Non-resuscitated Myocardial Infarction: diagnostic analysis of platelet function of a matched historical cohort of the ATLANTIS-ACS trial
  diagnostic analysis of platelet function: analysis of platelet aggregation using optical measurements
- Resuscitated Myocardial Infarction: diagnostic analysis of platelet function of the patient cohort included according to the inclusion criteria
  diagnostic analysis of platelet function: analysis of platelet aggregation using optical measurements
Arm/Group | Non-resuscitated Myocardial Infarction | Resuscitated Myocardial Infarction
Number analyzed (Participants) | 77 | 22
AU*min | 109 [73 to 182] | 253.8 [122.7 to 352.2]

2. Secondary Outcome: Number of Participants With Cumulative Clinical Endpoint of Death and Stent Thrombosis
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Non-resuscitated Myocardial Infarction | Resuscitated Myocardial Infarction
Number analyzed (Participants) | 77 | 22
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- Resuscitated MI: Death within the Observation period of 7 days; n=3
- Non Resuscitated MI: Death within the Observation period of 7 days; n=0
Arm/Group | Resuscitated MI | Non Resuscitated MI
All-Cause Mortality (participants affected / at risk) | 3/22 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/77
Other Adverse Events (participants affected / at risk) | 0/22 | 0/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resuscitated MI (N=22) | Non Resuscitated MI (N=77)
High on aspirin platelet reactivity (Blood and lymphatic system disorders) | 0 | NA — High on aspirin platele reactivity defined as collagene AUC > 500

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes